CLINICAL TRIAL: NCT06701357
Title: A Prospective, Open-label Phase II Study of Chidamide Plus R-CHOP + X in Previously Untreated Diffuse Large B-cell Lymphoma with Double Expression of MYC and BCL2.
Brief Title: CR-CHOP+X in Previously Untreated DEL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Principal Investigator, Ruijin Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-B41
Record Dates: First submitted 2024-11-21; First posted 2024-11-22 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: DLBCL
Keywords: DLBCL; double-expression; chidamide
MeSH Terms: interventions — orelabrutinib; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cluster1 DEL：CR-CHOP+PD1 inhibitor (Experimental): Participants who met the inclusion/exclusion criteria signed informed consent and received 1 course of CR-CHOP, followed by stratification of the remaining 5 cycles based on genetic subtypes. C1 plus PD1 inhibitor.
  Interventions: Drug: CR-CHOP+PD1 inhibitor
- Cluster 2 and 3 DEL：CR-CHOP plus Orelabrutinib (Experimental): Participants who met the inclusion/exclusion criteria signed informed consent and received 1 course of CR-CHOP, followed by stratification of the remaining 5 cycles based on genetic subtypes. C2 and C3 were treated with Orelabrutinib.
  Interventions: Drug: CR-CHOP + Orelabrutinib
- Tp53 mut DEL：CR-CHOP plus Decitabine (Experimental): Participants who met the inclusion/exclusion criteria signed informed consent and received 1 course of CR-CHOP, followed by stratification of the remaining 5 cycles based on genetic subtypes.TP53mut plus decitabine.
  Interventions: Drug: CR-CHOP + decitabine

INTERVENTIONS:
Drug: CR-CHOP+PD1 inhibitor — Rituximab 375 mg/m2 D1； Cyclophosphamide 750mg/m2 D2； Doxorubicin 50mg/m2 D2； Vincristine 1.4 mg/m2 D2； Prednisone 60 mg/m2 D2-6； Chidamide 20mg/d D1,4,8,11； PD1 200mg D1
  Arms: Cluster1 DEL：CR-CHOP+PD1 inhibitor
Drug: CR-CHOP + Orelabrutinib — Rituximab 375 mg/m2 D1； Cyclophosphamide 750mg/m2 D2； Doxorubicin 50mg/m2 D2； Vincristine 1.4 mg/m2 D2； Prednisone 60 mg/m2 D2-6； Chidamide 20mg/d D1,4,8,11； Orelabrutinib 150mg/qd D1-21
  Arms: Cluster 2 and 3 DEL：CR-CHOP plus Orelabrutinib
Drug: CR-CHOP + decitabine — Rituximab 375 mg/m2 D1； Cyclophosphamide 750mg/m2 D2； Doxorubicin 50mg/m2 D2； Vincristine 1.4 mg/m2 D2； Prednisone 60 mg/m2 D2-6； Chidamide 20mg/d D1,4,8,11； Decitabine 10mg/m2 D-5 - -1
  Arms: Tp53 mut DEL：CR-CHOP plus Decitabine

SUMMARY:
This is a prospective, single-arm, open-label phase II clinical trial that evaluates the efficacy and safety of CR-CHOP regimen combined with different targeted drugs based on different molecular subtypes in newly diagnosed DEL patients.

DETAILED DESCRIPTION:
Participants who met the inclusion/exclusion criteria signed informed consent and received 1 course of CR-CHOP, followed by stratification of the remaining 5 cycles based on genetic subtypes. C1 plus PD1 inhibitor; C2 and C3 were treated with orelabrutinib. TP53mut plus decitabine. During chemotherapy, routine evaluation was performed after each course of treatment, and an objective comprehensive evaluation of efficacy was performed after 3 courses of treatment. Efficacy evaluation Patients with CR or PR should continue the original treatment, and patients with SD or PD should be recommended second-line salvage treatment. For the first summary evaluation after completion of all treatments, CR patients are placed on chidamide maintenance therapy (2 years recommended unless intolerable toxicity or disease progression occurs).

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically confirmed diffuse large B-cell lymphoma with CD20 positive;
* 2. MYC and BCL2 are expressed simultaneously, WHO immunohistochemical standards: MYC≥40%, BCL2 ≥50%;
* 3. Age ≥ 18 years old, ≦75 years old;
* 4. ECOG physical status score of 0, 1 or 2;
* 5. No previous history of malignant tumors; No other tumors occurred simultaneously;
* 6. Patients judged by the investigator to have a life expectancy of at least 6 months;
* 7. The patient or his legal representative must provide written informed consent prior to any research special examination or procedure;
* 8. International prognostic Index (IPI) >1 score.

Exclusion Criteria:

* 1. Have previously received systemic or local treatment including chemotherapy;
* 2. Previously received autologous stem cell transplantation;
* 3. Previous history of other malignant tumors, except skin basal cell carcinoma and cervical carcinoma in situ;
* 4. Accompanied by uncontrolled cardiovascular and cerebrovascular diseases, coagulation disorders, connective tissue diseases, serious infectious diseases and other diseases;
* 5. Primary central nervous system lymphoma;
* 6. Left ventricular ejection fraction ≤ 50%;
* 7. Laboratory test values at the time of screening (unless due to lymphoma): A. Neutrophils <1.5*109/L; B. Platelet <75*109/L; C. ALT or AST were 2 times higher than the upper limit of normal, AKP and bilirubin were 1.5 times higher than the upper limit of normal; D. Creatinine levels higher than 1.5 times the upper limit of normal;
* 8. Other concurrent and uncontrolled medical conditions that the investigator believes will affect patient participation in the study;
* 9. Patients with mental illness or other patients known or suspected to be unable to fully comply with the study protocol;
* 10. Pregnant or lactating women;
* 11. People living with HIV;
* 12. Patients with positive HbsAg test results need to undergo HBV DNA test, and can be enrolled before turning negative. In addition, if the HBsAg test result is negative, but the HBcAb test is positive (regardless of the HBsAb status), HBV DNA test should also be performed. If the result is positive, the treatment should also be negative before admission.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
CRR（Complete response rate） | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=21 days]
  CR rate at the end of treatment by FDG-PET defined as the proportion of participants with CR at the end of treatment according to the 2014 Lugano Response Criteria; as determined by the investigator

SECONDARY OUTCOMES:
PFS（Progression-free survival） | 2-year
  PFS, defined as the time from treatment to the first occurrence of disease progression or relapse using the 2014 Lugano Response Criteria or death due to any cause, whichever occurs first; as determined by the investigator
OS（Overall survival） | 2-year
  OS defined as the time from treatment to death from any cause
ORR（Overall response rate） | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=21 days]
  ORR at treatment completion or discontinuation defined as the proportion of participants with partial response (PR) or CR at the end of treatment according to the 2014 Lugano Response Criteria; as determined by the investigator

CONTACTS AND LOCATIONS:
Locations (1):
- No. 197 Ruijin 2nd Road, Huangpu District, Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No